CLINICAL TRIAL: NCT07059403
Title: A Phase I, Randomized, Double Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability and Immunogenicity of SN2001 in Healthy Adult Subjects
Brief Title: A Study of SN2001 Dose, Safety & Immunogenicity in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chimivac INC (Industry)
Responsible Party: Sponsor
Organization: Chimigen Biomedical (Chengdu) Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMG.2001.101
Record Dates: First submitted 2025-06-20; First posted 2025-07-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B Infection
Keywords: SN2001; Chronic hepatitis B infection (CHB); Hepatitis B infection (HBV); Healthy Adult Subjects
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Participants will be randomized in a 3:1 ratio to receive 4 doses of either SN2001 or placebo.
  Interventions: Biological: SN2001
- Cohort B (Experimental): Participants will be randomized in a 3:1 ratio to receive 4 doses of either SN2001 or placebo.
  Interventions: Biological: SN2001
- Cohort C (Experimental): Participants will be randomized in a 3:1 ratio to receive 4 doses of either SN2001 or placebo.
  Interventions: Biological: SN2001

INTERVENTIONS:
Biological: SN2001 — 100 µg, for subcutaneous (SC) injection
  Other Names: Placebo
  Arms: Cohort A
Biological: SN2001 — 200 µg, for subcutaneous (SC) injection
  Other Names: Placebo
  Arms: Cohort B
Biological: SN2001 — 300 µg, for subcutaneous (SC) injection
  Other Names: Placebo
  Arms: Cohort C

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-ascending-dose study of SN2001 in healthy adult subjects. The study is designed to evaluate the safety, tolerability and immunogenicity of SN2001.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years, inclusive.
2. Body mass index (BMI) ≥18.0 kg/m2 and ≤ 32.0 kg/m2.
3. Participants are in good general health as determined by the investigator, based on a medical evaluation including medical history, vital signs, physical examination, 12-lead electrocardiogram, clinical laboratory tests.
4. Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as hysterectomy, bilateral ovariectomy or post-menopause. A postmenopausal state should be confirmed by at least 12 months since last menstrual period and FSH > 40 IU.
5. Women of childbearing potential (WOCBP) may be enrolled in the study if the participant:

   * has practiced highly-effective contraception for 28 days prior to first injection, and
   * has a negative pregnancy test at Screening, and
   * agrees to refrain from ova donation from Screening until 48 weeks after completion of the final injection, and
   * practices abstinence as part of her usual and preferred lifestyle, and
   * has agreed to continue highly-effective contraception from Screening until 48 weeks after completion of the final injection.
6. Male participants:

   * with documented bilateral orchiectomy, or
   * agrees to practice abstinence from penile-vaginal intercourse or use condoms from Screening until 48 weeks after completion of the final subcutaneous injection, and
   * agrees to refrain from sperm donation from Screening until 48 weeks after completion of the final injection, and
   * the highly effective contraceptive methods listed above should also apply to WOCBP partners of male participants for the specified duration, in addition to male condom use, from Screening until 48 weeks after completion of the final injection.
7. Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

1. History of Hepatitis B virus (HBV) infection as evidenced by detection of HBV Surface and Core antigens.
2. Clinical laboratory evidence of active infection with human immunodeficiency virus (HIV) infection, or hepatitis C virus (HCV) infection, or hepatitis A virus (HAV), or hepatitis D virus (HDV), or syphilis and/or any other chronic viral infection.
3. Known exposure (e.g., sexual contact or blood exposure) to HBV within the past 6 weeks.
4. History of HBV vaccination:

   * Have not previously been vaccinated in the community for Hepatitis B (Engerix-B or similar), or
   * Have received any HBV vaccination (documented evidence of vaccination, or verbal history of vaccination) and a seroprotective Hepatitis B surface antibody (HBsAb) titre <10 milli-international units per milliliter (mIU/mL) at screening, or
   * Have received any HBV vaccination (documented evidence of vaccination, or verbal history of vaccination) within 6 months prior to the screening visit, or
   * Have HBV vaccination scheduled plan within 48 weeks after the final study drug dosing.
5. Receipt of any investigational drug or vaccine or medical device clinical trial within 3 months or 5 half-lives (whichever is greater) prior to screening.
6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin greater than or equal to 1.5×ULN, or any other laboratory values considered clinically significant abnormalities and unacceptable by the Investigator at screening.
7. Current or a history of any clinically significant medical illness or medical disorders the investigator considers should exclude including (but not limited to) neurological disease, cardiovascular disease, hepatic or renal disease (such as chronic liver disease), gastrointestinal tract disease, respiratory disease, metabolism, skeletal system diseases or other conditions known to put the subject at significant risk.
8. History of Cancer within 3 years, excluding basal cell carcinoma, squamous cell carcinoma, or cervical intraepithelial neoplasia, which is cured is allowed.
9. Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus.
10. History of any severe trauma or major surgical condition within 3 months or planned to undergo surgery during the study period.
11. Presently receiving (or history of receiving), during the preceding 3 months or 5 half-lives (whichever is greater), any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable). Inhaled and topical corticosteroids, intranasal corticosteroids (e.g. Nasonex for allergic rhinitis) are allowed.
12. Used prescription drugs or vaccines within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug.
13. Used over-the-counter (OTC) medication or herbal supplements, excluding routine vitamins, within 7 days before the first dose of study drug, unless determined by the Investigator and the Sponsor to be not clinically relevant and unlikely to impact on study outcomes. Paracetamol or ibuprofen can be considered an exception for the treatment of headaches or any other pain for eligibility purposes.
14. Participants smoke ≥ 10 cigarettes a day within 3 months before screening, or those who cannot stop using any tobacco products from screening until 24 weeks after the final injection.
15. History or clinical evidence of alcohol abuse, within the 3 months before screening, and unwillingness to abstain from alcohol within 3 weeks after the final study drug dosing. Alcohol abuse is defined as regular weekly intake of more than 14 units for male and 10 units for female (unit: 1 glass of wine [125 mL] = 1 measure of spirits = ½ pint of beer).
16. History or clinical evidence of drug abuse, within the 12 months before screening. Drug abuse is defined as compulsive, repetitive, and/or chronic use of drugs or other substances with or without problems related to their use and/or were stopping or a reduction in dose will lead to withdrawal symptoms.
17. Confirmed positive results from drug of abuse (amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, phencyclidine, tetrahydrocannabinol, cotinine, tricyclic anti-depressants) or from the alcohol breath test at screening.
18. History of significant local or systemic reactogenicity (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration).
19. Donated more than 400 mL of blood within 30 days before the first dose of study drug.
20. Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | from the time of the first study injection through 48 Weeks after the final study injection
  Number of subjects with AEs assessed by the 2007 FDA Guidance to Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
  Solicited local injection site reactions and solicited systemic symptoms on the day of each study injection and for 7 days.
  Non-serious unsolicited AEs will be collected until 21 days after 1st, 2nd, and 3rd study injection, and until 28 days after last study injection.
  All serious adverse events (SAEs), medically attended adverse events (MAAEs) and adverse events of special interest (AESIs) must be collected from the time of the first study injection through 48 weeks after the final study injection.
Number of subjects with clinically significant abnormalities in vital signs graded by 2007 FDA Guidance. | from the time of the first study injection through 48 Weeks after the final study injection
  Vital sign measurements include blood pressure, pulse rate, respiratory rate and temperature.
  The number (n) and percentages (%) of "normal", "abnormal not clinically significant (NCS)", and "abnormal clinically significant (CS)" from baseline through the worst post-baseline visit will be summarized.
Number of subjects with clinically significant abnormalities in physical examination graded by 2007 FDA Guidance. | from the time of the first study injection through 48 Weeks after the final study injection
  A full physical examination will include general appearance, head, neck, chest/respiratory, heart/cardiovascular, gastrointestinal/liver, extremities, skin, and neurological assessments.
  The number (n) and percentages (%) of "normal", "abnormal not clinically significant (NCS)", and "abnormal clinically significant (CS)" from baseline through the worst post-baseline visit will be summarized.
Number of subjects with clinically significant abnormalities in 12-lead electrocardiogram (ECG) graded by 2007 FDA Guidance. | from the time of the first study injection through 48 Weeks after the final study injection
  12-lead ECGs will include heart rate, PR intervals, QRS intervals, QT intervals, and QTcF intervals.
  The number (n) and percentages (%) of "normal", "abnormal not clinically significant (NCS)", and "abnormal clinically significant (CS)" from baseline through the worst post-baseline visit will be summarized.
Number of subjects with clinically significant abnormalities in laboratory parameters graded by 2007 FDA Guidance. | from the time of the first study injection through 48 Weeks after the final study injection
  Laboratory parameters will include hematology, chemistry, coagulation parameters, urinalysis, etc.
  The number (n) and percentages (%) of "normal", "abnormal not clinically significant (NCS)", and "abnormal clinically significant (CS)" from baseline through the worst post-baseline visit will be summarized in all parameters.
  Mean change and shift from baseline to each scheduled post-baseline visit will be summarized in all quantitative parameters.

SECONDARY OUTCOMES:
Serum SN2001 antibody titers. | from before the first study injection through 24 Weeks after the final study injection
  Serum SN2001 antibody titers will be measured by enzyme linked immunosorbent assay (ELISA).
  Geometric mean titers (GMTs), and 95% confidence intervals (95% CI) will be calculated per cohort.
Seroconversion (SN2001). | from before the first study injection through 24 Weeks after the final study injection
  Serum SN2001 antibody titers will be measured by ELISA. Seroconversion is defined as the appearance of antibodies [i.e., concentrations/titer greater than or equal to the lower limit of quantification (LLOQ)] in the serum of subjects seronegative before investigational product administration.
Serum HBV Core protein antibody titers. | from before the first study injection through 24 Weeks after the final study injection
  Serum HBV Core protein antibody titers will be measured by ELISA. Geometric mean titers (GMTs), and 95% confidence intervals (95% CI) will be calculated per cohort.
Seroconversion (HBV Core protein). | from before the first study injection through 24 Weeks after the final study injection
  Serum HBV Core protein antibody titers will be measured by ELISA. Seroconversion is defined as the appearance of antibodies (i.e., concentrations/titer greater than or equal to the LLOQ) in the serum of subjects seronegative before investigational product administration.
Serum HBV PreS1/S2 protein antibody titers. | from before the first study injection through 24 Weeks after the final study injection
  Serum HBV PreS1/S2 protein antibody titers will be measured by ELISA. Geometric mean titers (GMTs), and 95% confidence intervals (95% CI) will be calculated per cohort.
Seroconversion (HBV PreS1/S2 protein). | from before the first study injection through 24 Weeks after the final study injection
  Serum HBV PreS1/S2 protein antibody titers will be measured by ELISA. Seroconversion is defined as the appearance of antibodies (i.e., concentrations/titer greater than or equal to the LLOQ) in the serum of subjects seronegative before investigational product administration.
Frequency of HBV core-specific IFN-γ-secreting peripheral blood mononuclear cells (PBMCs). | from before the first study injection through 24 Weeks after the final study injection
  HBV core-specific IFN-γ-secreting PBMCs is measured by immunosorbent spot (ELISpot) assay. Frequency of HBV core-specific IFN-γ-secreting PBMCs is expressed as HBV core-specific T-cells per million peripheral blood mononuclear cells (HBV core-specific IFN-γ-secreting PBMCs /million PBMCs).
Frequency of HBV core-specific IL-4-secreting peripheral blood mononuclear cells (PBMCs). | from before the first study injection through 24 Weeks after the final study injection
  HBV core-specific IL-4-secreting PBMCs is measured by immunosorbent spot (ELISpot) assay. Frequency of HBV core-specific IL-4-secreting PBMCs is expressed as HBV core-specific T-cells per million peripheral blood mononuclear cells (HBV core-specific IL-4-secreting PBMCs /million PBMCs).

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Ltd., Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No